CLINICAL TRIAL: NCT02537613
Title: A Phase Ib Study of Ibrutinib in Combination With Obinutuzumab in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: A Study of Ibrutinib + Obinutuzumab in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Matthew S. Davids, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-283
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A- obinutuzumab -> ibrutinib (Experimental): Participants enrolled in Arm A will receive obinutuzumab weekly starting cycle 1, and will receive obinutuzumab monthly during cycles 2-6. Participants will begin to take ibrutinib daily starting cycle 2 and will continue with daily ibrutinib until the end of treatment.
  Interventions: Drug: Obinutuzumab; Drug: Ibrutinib
- Arm B- ibrutinib -> obinutuzumab (Experimental): Participants enrolled in Arm B will begin to take ibrutinib daily starting cycle 1 and will continue with daily ibrutinib until the end of treatment. Participants will begin to receive obinutuzumab weekly starting cycle 2, and will receive obinutuzumab monthly during cycles 3-7
  Interventions: Drug: Obinutuzumab; Drug: Ibrutinib
- Arm C- obinutuzumab/ibrutinib (Experimental): Participants enrolled in Arm C will begin to take ibrutinib daily starting cycle 1 and will continue with daily ibrutinib until the end of treatment. At the same time, participants will begin to receive obinutuzumab weekly starting cycle 1, and will receive obinutuzumab monthly during cycles 2-6.
  Interventions: Drug: Obinutuzumab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab given weekly during cycle 1, then monthly during cycles 2-6
  Other Names: Gazyva; GA-101
Drug: Ibrutinib — Ibrutinib given once daily by mouth
  Other Names: Imbruvica

SUMMARY:
This research study is evaluating a combination of two drugs, ibrutinib and obinutuzumab, as a possible treatment for Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the best order of administration of these two drugs. "Investigational" means that the intervention is being studied. The FDA (the U.S. Food and Drug Administration) has approved ibrutinib and obinutuzumab individually for the treatment of patients with Chronic Lymphocytic Leukemia, your type of cancer. However, the FDA has not approved the combination of these two drugs as a treatment for any disease.

Ibrutinib is a type of drug called a kinase inhibitor. It is believed to block a type of protein called a kinase that helps leukemia cells live and grow. By blocking this, it is possible that the study drug will kill cancer cells or stop them from growing.

Obinutuzumab is a type of drug called a monoclonal antibody. It is believed to attach to a protein called CD20 on the outside of a Chronic Lymphocytic Leukemia cell. By attaching to the cell, the antibody can cause the Chronic Lymphocytic Leukemia cell to die.

In this research study, the investigators are assessing the safety of various dosing regimens of ibrutinib and obinutuzumab. The investigators are trying to determine whether it is better to give one drug before the other or if they can be started at the same time.

ELIGIBILITY:
Inclusion criteria:

* Must have a confirmed diagnosis of Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma as per IW-CLL 2008 criteria and require therapy based on meeting at least one of the following criteria:

  * Evidence of progressive marrow failure with anemia (hemoglobin <11.0 g/L) and/or thrombocytopenia (platelets <100 x 10^9/L)
  * Massive (≥6 cm below the left costal margin), progressive, or symptomatic splenomegaly
  * Massive nodes (at least 10 cm longest diameter), progressive, or symptomatic lymphadenopathy
  * Progressive lymphocytosis with an increase of more than 50% over a 2-month period or LDT of <6 months.
  * Autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids
  * Constitutional symptoms, defined as 1 or more of the following:

    * unintentional weight loss >10% within 6 months prior to screening
    * significant fatigue (inability to work or perform usual activities) fevers >100.5° F or 38.0° C for 2 or more weeks prior to screening without evidence of infection
    * night sweats for more than 1 month prior to screening without evidence of infection
* Relapsed after or refractory to at least one prior Chronic Lymphocytic Leukemia-directed therapy
* Age greater than or equal to 18 years
* ECOG Performance Status <2
* Heme criteria at screening, unless significant bone marrow involvement of Chronic Lymphocytic Leukemia confirmed on biopsy:

  * Absolute Neutrophil Count (ANC) ≥500 cells/mm3 (0.5 x 10^9/L). Growth factor allowed to achieve
  * Platelet count ≥25,000 cells/mm3 (25 x 10^9/L) independent of transfusion within 7 days of screening
* Adequate hepatic function defined as: AST and ALT ≤ 4.0 x upper limit of normal (ULN), bilirubin ≤2.0 x upper limit of normal (ULN) unless bilirubin rise is due to Gilbert's syndrome)
* Adequate renal function defined by serum creatinine <2.0 x upper limit of normal (ULN) unless due to biopsy proven Chronic Lymphocytic Leukemia kidney infiltration
* Women of child-bearing potential and men must agree to use adequate contraception
* Patients who have undergone prior allo transplant are eligible provided that their transplant day 0 is > 6 months from their first dose of study drug

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Prior treatment with either obinutuzumab or ibrutinib
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for ≥3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
  * Low-risk prostate cancer on active surveillance
* Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc., or chronic administration of >20 mg/day of prednisone) within 28 days of the first dose of study drug.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Recent infection requiring systemic treatment that was completed ≤7 days before the first dose of study drug.
* Known bleeding disorders or hemophilia.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Known history of HIV or active hepatitis C virus (HCV) or hepatitis B virus (HBV).
* Any uncontrolled active systemic infection.
* Major surgery within 4 weeks of first dose of study drug.
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 CHF as defined by the NYHA Functional Classification; or a history of Myocardial Infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
* Lactating or pregnant.
* Patients receiving any other study agents
* Patients with known Central Nervous System involvement
* Baseline QT Interval Corrected by the Fridericia Correction Formula (QTcF) >480 ms unless Left Bundle Branch Block
* Patients who require warfarin or other vitamin K antagonists for anticoagulation
* Concurrent administration of strong inhibitors or inducers of CYP3A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Baseline to 6 Months
  To assess the safety of 3 different dosing regimens of ibrutinib plus obinutuzumab in patients with relapsed/refractory CLL

SECONDARY OUTCOMES:
Overall Response Rate | 6 Months
  To assess the efficacy of ibrutinib plus obinutuzumab in patients with relapsed/refractory CLL as measured by:
Partial Response Rate | 6 Months
  To assess the efficacy of ibrutinib plus obinutuzumab in patients with relapsed/refractory CLL as measured by:
Complete Response Rate | 6 Months
  To assess the efficacy of ibrutinib plus obinutuzumab in patients with relapsed/refractory CLL as measured by:
Minimal residual disease (MRD) status in the bone marrow and blood | 6 Months
  To assess the efficacy of ibrutinib plus obinutuzumab in patients with relapsed/refractory CLL as measured by:
Duration of Response | 2 Years
  To assess the efficacy of ibrutinib plus obinutuzumab in patients with relapsed/refractory CLL as measured by:
Progression Free Survival | 2 Years
  To assess the efficacy of ibrutinib plus obinutuzumab in patients with relapsed/refractory CLL as measured by:
Overall Response Rate | 2 Years
  To assess the efficacy of ibrutinib plus obinutuzumab in patients with relapsed/refractory CLL as measured by:

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davids, MD, MMSc, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Rochester Wilmot Cancer Inst., Rochester, New York
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No